CLINICAL TRIAL: NCT05344131
Title: Investigation of the Effectiveness of a Biopsychosocial-Based Exercise Model in Rheumatic Diseases: A Mixed Methods Research With Patients' Perspectives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nazli Elif Nacar, Physiotherapist (MSc), Kahramanmaras Sutcu Imam University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kahramanmaras SIU
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Rheumatic Diseases
Keywords: Biopsychosocial Model; Rheumatic diseases; Qualitative Research; Exercise
MeSH Terms: conditions — Rheumatic Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The quantitative part of the study (BETY exercise group) (Experimental): intervention group Bilişsel Egzersiz Terapi Yaklaşımı (BETY, Cognitive Exercise Therapy Approach) is a group exercise method that conforms to the biopsychosocial model.
  Exercise dosage is 60 minute three days a week.
  Interventions: Other: Bilişsel Egzersiz Terapi Yaklaşımı (BETY, Cognitive Exercise Therapy Approach)
- The quantitative part of the study (Control group) (No Intervention): Control group No intervention
- The qualitative part of the study (Experimental): Regularly participated in the BETY program for at least one year Bilişsel Egzersiz Terapi Yaklaşımı (BETY, Cognitive Exercise Therapy Approach) is a group exercise method that conforms to the biopsychosocial model.
  Exercise dosage is 60 minute three days a week.
  Interventions: Other: Bilişsel Egzersiz Terapi Yaklaşımı (BETY, Cognitive Exercise Therapy Approach)

INTERVENTIONS:
Other: Bilişsel Egzersiz Terapi Yaklaşımı (BETY, Cognitive Exercise Therapy Approach) — Biopsychosocial approach
  Arms: The qualitative part of the study; The quantitative part of the study (BETY exercise group)

SUMMARY:
Biopsychosocial approaches are recommended in rheumatic diseases. Because the nature of these diseases is based on the person's ability to cope with their chronic disease. Moreover, rheumatic diseases, which are included in chronic diseases; It creates a comprehensive picture with loss of function, fatigue, insomnia, sexual reluctance, negative mood, social isolation and persistent pain accompanying them. This picture requires comprehensive treatments to include the symptoms. For this reason, biopsychosocial models are drawing attention day by day and it is underlined that a holistic approach to rheumatic patients is necessary. For all these negative conditions, exercise offers treatment as an important parameter. However, it seems that no named, exercise-based biopsychosocial models recommended for rheumatic diseases have been encountered. Studies show that cognitive behavioral therapies play a role when it is necessary to approach this patient group holistically. Patients diagnosed with rheumatism, who have applied to Hacettepe University Faculty of Health Sciences Physiotherapy and Rehabilitation Department since 2004, were included in group training where they could do clinical pilates exercises. Dance therapy-authentic movement was added to the exercise program in order to break the physiological connection of the vicious circle between the awareness gained in 2009 and the pain and anxiety. In 2010, the relationship between anxiety and pain led to the addition of knowledge management in sexuality this time. It was published in the form of a rheumatism book in 2014. In 2015, BETY received trademark registration. In this process, the patients learned to manage their inflammatory pain during the day by applying the pain management strategy individually. The exercise program, which was applied for one hour 3 days a week, was created by applying scales for the diagnosis of diseases during the evaluation phase.However, the patients stated that the relevant scales did not show the change in themselves, and that they experienced different changes. During this period, patients were asked to form sentences expressing the characteristics of change. The sentences formed were simplified by removing the same ones. These sentences were tested on rheumatic patients who did not participate in the BETY group. The item pool was formed by making additions related to activities of daily living. The draft was sent to rheumatologists and their opinions were taken. The opinions of the rheumatologists were shared with the patients, and the final version of the items was given in 2017. This scale was started to be applied to individuals with rheumatism who participated in the BETY program. It was also used for evaluation purposes for patients who did not participate in the exercise group but were given a home program after only the first interview. In this process, which formed the basis for the development of a scale, a qualitative study was needed that investigated the recovery characteristics of the patients and the reasons for their persistence in exercise. This qualitative study aims to reveal in detail the change created by an exercise-based biopsychosocial model in patients with rheumatism. Putting all these mentioned processes in writing and presenting them to the literature will be the efficiency of this study.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed rheumatic diseases
* 18 years and over

Exclusion Criteria:

* presence of infection and fever, deformity that does not allow exercise, cardiopulmonary disorders, uncontrolled endocrine system diseases, and severe psychiatric illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Qualitative methods | after minimum one year participated BETY group
  We aimed to complete qualitative semi-structured interviews to investigate biopsychosocial perspectives of patients with rheumatic diseases in each arm of the study. Two pre-prepared interview topic guides were developed collaboratively by the research team with the project steering group which included lay members.
Quantitative methods - Assessment of biopsychosocial status Bilişsel Egzersiz Terapi Yaklaşımı-Biopsychosocial Questionnaire (BETY-BQ) | before -12 weeks after.
  The scale consists of 30 items. The scoring of the scale was made using a 5-point Likert system. Each question is scored as "No never: 0 Yes rarely: 1 Yes sometimes: 2 Yes often: 3 Yes always: 4" and gives a total score over 30 items. A high score means that the biopsychosocial situation is 'bad'.

SECONDARY OUTCOMES:
Quantitative methods - Assessment of functionality Health Assessment Questionnaire (HAQ) | before -12 weeks after.
  The functional status of the patients was determined by the Health Assessment Questionnaire. The 20-question scale has 8 subtitles that include dressing, sitting, eating, walking, hygiene, reaching out, grasping, and daily life activities. Each answer is scored between 0 and 3 points. It means "0 = Without difficulty, 1 = A little difficult, 2 = Very difficult and 3 = I can never do it". The total score is the average score derived from 8 points for each category.High score indicates low functional status.
Quantitative methods - Assessment of emotional status Hospital Anxiety and Depression Scale (HADS) | before -12 weeks after.
  The anxiety and depression of the patients was determined by Hospital Anxiety and Depression Scale (HADS). This questionnaire is consisting of 14 questions with 4 options. The higher the score, the higher the anxiety and depression levels.
Quantitative methods - Assessment of quality of life Short Form 36 Health Survey Questionnaire (SF-36) | before -12 weeks after.
  The quality of life of the patients was evaluated with the SF-36 scale. Separate scores are obtained for each sub-parameter and scores range from 0-100. 100 points indicate good health, 0 points indicate poor health

CONTACTS AND LOCATIONS:
Overall Officials: EDİBE Unal, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)